CLINICAL TRIAL: NCT06054789
Title: Clinical Study on 68Ga-PSMA-33 for PET/CT Imaging of Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, FengWang, Professor, Nanjing First Hospital, Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 68Ga-PSMA-33
Record Dates: First submitted 2023-09-12; First posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Prostate Cancer
Keywords: Prostate-Specific Membrane Antigen (PSMA); PET/CT; Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-PSMA-33 (Experimental): For the injection, subjects will receive a target dose of 3-7mCi 68Ga-PSMA-33 as a bolus injection. Among them, 3~4 subjects will additionally inject with 68Ga-PSMA-617 (3-7mCi).
  Interventions: Drug: 68Ga-PSMA-33

INTERVENTIONS:
Drug: 68Ga-PSMA-33 — Subjects will receive one injection of 68Ga-PSMA-33/PSMA-617 (3-7mCi ), a PET radiopharmaceutical selective for Prostate-Specific Membrane Antigen. 68Ga-PSMA-33/PSMA-617 injection will be followed by a 10 ml saline flush.
  Other Names: 68Ga-PSMA-617

SUMMARY:
The purpose of this study is to determine the pharmacokinetics, dosimetry, tolerance, tumor detection rate of 68Ga-PSMA-33 in patient with Prostate Cancer (PCa).

DETAILED DESCRIPTION:
This study is design to prospectively investigate the safety and efficacy of 68Ga-PSMA-33 in the early diagnosis of Prostate Cancer (PCa). The specific objectives are the determination of pharmacokinetics, dosimetry, tolerance and tumor detection rate of 68Ga-PSMA-33 in patient with PCa. While PSMA is expressed at low levels in normal prostate epithelium, it is overexpressed (up to 1000 times higher) in 90-95% of prostate cancers, make PSMA an attractive target for the diagnosis and treatment of PCa. 68Ga-PSMA-33 as a new PSMA targeted probe was prepared and showed good uptake on PCa cell line and animal studies.

The study intends to recruit 8 PCa volunteers to participate in the experiment. All patients were intravenously injected with 68Ga-PSMA-33 and underwent PET/CT at 0.5, 1, 2 and 4 h, respectively. For comparison, 3 patients were additionally received 68Ga-PSMA-617 PET/CT imaging. The images were interpreted by two experienced physician and the SUVmax or SUVmean of physiological organs and tumor lesions were collected.

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* Age 18 years or older
* Patients must have histologically or cytologically confirmed localized or metastatic prostate cancer
* Creatinine less than or equal to 1.5 X upper limit of normal
* ECOG performance status 0 - 2, inclusive
* Able to tolerate the physical/logistical requirements of a PET/CT scan including lying supine (or prone) for up to 30 minutes and tolerating intravenous cannulation Patient with complete clinical data.
* The effects of 68Ga-PSMA-33 on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.
* Able to understand and provide written informed consent

Exclusion Criteria:

* Patient age < 18 years
* Received radioisotope diagnosis or treatment before enrollment, and the time window did not exceed 10 physical half-lives
* Malignancy other than current disease under study
* Patient simultaneously participating in another clinical trial
* Patient who cannot stay on PET/CT
* Patient with HIV, HCV, HVB infection or other serious chronic infection
* Patient with liver and kidney function (GFR less than 50 ml/min) disease
* Cannot receive furosemide, allergy to sulfa or sulfa-containing medications
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Tumor detection rate | 2 years
  Comparing the number of tumor detected by 68Ga-PSMA-33 and 68Ga-PSMA-617 PET/CT.
Standardized uptake value (SUV) of tumor | 2 years
  Comparing the SUVmax of tumor derived from 68Ga-PSMA-33 and 68Ga-PSMA-617 PET/CT.

SECONDARY OUTCOMES:
Safety and Tolerability Profile Measured by Adverse Events (AEs) | 2 years
  Safety and tolerability profile for the administration of 68Ga-PSMA-33 and positron emission tomography (PET) scanning are measured by number of participants with adverse events (AEs).

CONTACTS AND LOCATIONS:
Overall Officials: Feng Wang, Study Director — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- 68Ga-PSMA-33 PET/CT imaging, Nanjing, Jiangsu, China